CLINICAL TRIAL: NCT05833607
Title: Effects of Systemic Blood Pressure Targets on Cerebral Hemodynamics in Septic Shock: a Prospective Study
Brief Title: Effects of Targets of Blood Pressure on Cerebral Hemodynamics in Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Other Study IDs: 28134720.1.0000.0048
Record Dates: First submitted 2023-03-29; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Septic Shock; Cerebral Autoregulation
Keywords: Septic Shock; Cerebral autoregulation; Cerebral hemodynamics
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALL PATIENTS: All patients are monitored with the transcranial Doppler helmet and the 2Hz probe in one of the middle cerebral hemispheres and the Brain 4 care on the other side.
  Necessary monitoring: arterial line, electrocardiographic monitor, pulse oximetry, temperature. ETCO2 monitoring whenever possible.
  Step 1: Test arterial line circuit, ensure proper temperature, arterial blood gases Step 2: Record data with the patient's baseline pressure (data from the monitor, transcranial doppler and brain4care), for 5 min Step 3: Vasopressor titrant for 3 MAP targets (65, 75 and 85 mmHg) , record data with the patient's baseline pressure (data from the monitor, transcranial doppler and brain4care), each target record for 3 minutes Step 4: Arterial blood gases, gradually restore PAM to baseline value

SUMMARY:
The sudy objective is to evaluate the cerebral haemodynamic status in different ranges of systemic arterial pressure in patients with septic shock by noninvasive tools, transcranial doppler and intracranial compliance by mechanical sensor (B4C).

Patients participating in the study will be submitted to different levels of arterial pressure, titrated with vasopressor and them their cerebral hemodynamic variables will be evaluated,

DETAILED DESCRIPTION:
Sepsis is the most prevalent cause of admissions to the intensive care unit (ICU) and many of these patients develop septic shock (SC) (need for vasoactive drug, after adequate fluid administration, plus hyperlactatemia). The SC involvement is systemic, so the investigators started to monitor organ dysfunctions and their perfusion windows, including neurological disorders, when is affected, in addition to indicating severity, are also a predictor of worse prognosis.

The principle of cerebral autoregulation (CA) is the basic defense mechanism against pressure oscillations in the most diverse contexts. The SC is a state of vasodilation and consequent drop in mean arterial pressure (MAP), that under normal physiological conditions would be compensated by CA. But it is not known exactly how CA performance at this profile of patients.

The investigators will assess cerebral hemodynamics in SC patients at different MAP targets, in order to identify whether this regulatory variable would be able to generate better parameters of cerebral hemodynamics.

Some smaller studies have shown that liver and heart dysfunction correlate with worsening autoregulation. Another clinical trial showed an inverse relationship between CA and the Sequential Organ Failure Assessment, in addition to the loss of CA in patients with circulatory shock in general. Post-mortem data found generalized ischemic lesions in the brain of septic patients, which translates into a state of reduction at vascular flow. This patient profile has more blood-brain barrier dysfunction, but further studies are needed to correlate CA and CS.

The study will be carried out in the ICU of Hospital São Rafael (HSR), located in the city of Salvador-Ba, Brazil. For the evaluation of cerebral hemodynamics Transcranial Doppler and a Mechanical sensor (B4C) will be used.

Data collection on admission will include the following: demographic characteristics, comorbidities, source of infection, Sequential Organ Failure Assessment (SOFA) at ICU admission, temperature, Glasgow Coma scale (GCE) or Richmond Agitation Sedation Scale (RASS), mechanical ventilation, arterial blood gasses before and after the protocol.

All patients will be monitored with an arterial line, cardioscopy, pulse oximetry and capnography (if unavailable at the time of collection, this will be described). Before starting the monitoring, the proper functioning of the arterial circuit will be confirmed and a blood gas analysis will be collected, as well as at the end.

The investigators will collet data with the patient's baseline pressure for 5 minutes (T0), then through the titration of vasopressors, for another 5 minutes each mean arterial pressure target at 65mmHg (T1), 75 mmHg (T2) and 85 mmHg (T3). After collection, the baseline mean arterial pressure will be restored

ELIGIBILITY:
Inclusion Criteria:

* < 48 hours in the intensive care unit
* Septic shock (sepsis 3.0)

Exclusion Criteria:

* No window for DTC
* Hepatic or uremic encephalopathy
* Pregnancy
* Acute or prior structural neurological insult
* Exogenous intoxication
* Dementia
* Chronic Obstructive Pulmonary Disease
* Instability for acute arrhythmia
* Extracorporeal support by modifying the pulse wave form (intra aortic balloon pump and Extracorporeal membrane oxygenation
* Extreme severity, with imminent risk of death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock with less than 48 hours of ICU stay
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-07 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate the effects of cerebral haemodynamic in patients with septic shock in different targets of MAP, through ARI (by Transcranial Doppler), and intracranial compliance by mechanical sensor (B4C) | Data will be obtained at the time of collection (mean arterial pressure targets) and subsequently analyzed
  This outcome will be analyzed by transcranial Doppler (ARI, PI) and B4C (intracranial compliance) index). Data will be obtained at the time of collection (mean arterial pressure targets) and subsequently analyzed

SECONDARY OUTCOMES:
Assess factors that influence cerebral autoregulation (by ARI) and intracranial compliance (B4C) | Data will be obtained at the time of collection (mean arterial pressure targets) and subsequently analyzed
  To verify clinical factors that influence cerebral autoregulation (CA) and intracranial compliance of septic patients
Evaluate the correlation between CA by TDC and B4C index. | Data will be obtained at the time of collection (mean arterial pressure targets) and subsequently analyzed
  Report the similarity between the two indices
Correlate mechanical ventilation time with perfusion pressure value | Mechanical ventilation time up to 28 days
  Observation that there is a correlation between the duration of mechanical ventilation and the patient's baseline perfusion pressure
Explore the correlation between incidence of brain dysfunction | Until 28º day
  Brain dysfunction will be considered as: Glasgow Coma Scale score < 15 or when disorientation, altered thinking or agitation was reported by the attending physician, independently of the use of sedatives/analgesics and in the absence of previous neurological diseases (i.e., dementia, cerebrovascular disease, brain tumors, previous traumatic brain injury) with DTC and B4C index.

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Caldas, Phd, Principal Investigator — D'Or Institute for Research and Education (IDOR), Hospital São Rafael; Pedro Cury, Study Chair — D'Or Institute for Research and Education (IDOR), Hospital São Rafael
Locations (1):
- São Rafael Hospital, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No
We don't have that plan, but if the data is useful for larger research, no problem.

REFERENCES:
- [Derived] Cury P, Passos RDH, Alves F, Brasil S, Frigieri G, Taccone FS, Panerai RB, Caldas J. Impact of different blood pressure targets on cerebral hemodynamics in septic shock: A prospective pilot study protocol-SEPSIS-BRAIN. PLoS One. 2024 Oct 14;19(10):e0304412. doi: 10.1371/journal.pone.0304412. eCollection 2024. PMID 39401208
- See also: The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3) — http://pubmed.ncbi.nlm.nih.gov/26903338/
- See also: Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021 — https://pubmed.ncbi.nlm.nih.gov/34599691/
- See also: Cerebral dysfunctions caused by sepsis during ageing — https://pubmed.ncbi.nlm.nih.gov/34764472/
- See also: Cerebral autoregulation — https://pubmed.ncbi.nlm.nih.gov/2201348/
- See also: Dynamic Autoregulation is Impaired in Circulatory Shock — https://pubmed.ncbi.nlm.nih.gov/31764617/
- See also: Impaired cerebral autoregulation is associated with brain dysfunction in patients with sepsis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6280405/
- See also: Waveform Morphology as a Surrogate for ICP Monitoring: A Comparison Between an Invasive and a Noninvasive Method — https://pubmed.ncbi.nlm.nih.gov/35332426/
- See also: Noninvasive intracranial pressure waveforms for estimation of intracranial hypertension and outcome prediction in acute brain-injured patients — https://link.springer.com/article/10.1007/s10877-022-00941-y
- See also: Persistent cognitive impairment, hippocampal atrophy and EEG changes in sepsis survivors — https://pubmed.ncbi.nlm.nih.gov/23134661/
- See also: POCUS, how can we include the brain? An overview — https://janesthanalgcritcare.biomedcentral.com/articles/10.1186/s44158-022-00082-3
- See also: A Novel Noninvasive Technique for Intracranial Pressure Waveform Monitoring in Critical Care — https://pubmed.ncbi.nlm.nih.gov/34945774/
- See also: Daily blood pressure variability in relation to neurological functional outcomes after acute ischemic stroke — https://www.frontiersin.org/articles/10.3389/fneur.2022.958166/full